CLINICAL TRIAL: NCT06531941
Title: An Extension Study to Evaluate the Long-Term Safety and Tolerability of MBX 2109 in Patients With Hypoparathyroidism Who Completed the 12-Week Treatment Period in the Phase 2 Study, MBX-2H1002 Study (Avail-Ext)
Brief Title: Extension Study to Evaluate the Long-Term Safety and Tolerability of MBX 2109 in Patients With Hypoparathyroidism
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MBX Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MBX-2H1004
Record Dates: First submitted 2024-07-16; First posted 2024-08-01 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroid; Hypopara; Thyroid; MBX 2109
MeSH Terms: conditions — Hypoparathyroidism; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 400 µg once-weekly by subcutaneous injection (Experimental)
  Interventions: Drug: 400 µg of MBX 2109 once-weekly by subcutaneous injection
- 200-1600 µg once-weekly by subcutaneous injection (Experimental)
  Interventions: Drug: 200-1600 µg of MBX 2109 once-weekly by subcutaneous injection

INTERVENTIONS:
Drug: 400 µg of MBX 2109 once-weekly by subcutaneous injection — Supplied as 1.5 mg per vial, to be reconstituted in 1.4 mL water for injection (diluent) to a concentration of 1.0 mg/mL.
  Patients who received Placebo in the Phase 2 MBX-2H1002 study, will initiate treatment with 400 µg subcutaneous MBX 2109 once-weekly
  Arms: 400 µg once-weekly by subcutaneous injection
Drug: 200-1600 µg of MBX 2109 once-weekly by subcutaneous injection — Supplied as 1.5 mg per vial, to be reconstituted in 1.4 mL water for injection (diluent) to a concentration of 1.0 mg/mL.
  Patients treated with MBX 2109 in the Phase 2 MBX-2H1002 study will continue at the screening visit in the extension study on the same dose they were receiving at the Week 11 Visit in Study MBX-2H1002.
  The maximum allowed dose is 1600 μg weekly administered subcutaneously in the abdomen, rotating injection sites. Doses of MBX 2109 study drug greater than 1000 μg will be administered subcutaneously in two separate, equal injections.
  Arms: 200-1600 µg once-weekly by subcutaneous injection

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of MBX 2109 in patients with hypoparathyroidism who completed the 12-week treatment period in the Phase 2 study, MBX-2H1002.

DETAILED DESCRIPTION:
This study is to investigate the long-term safety and tolerability of MBX 2109 administered once weekly to patients with hypoparathyroidism. Additionally, the ability of MBX 2109 to maintain serum calcium levels within the normal range without the need for active vitamin D and to reduce elemental calcium supplements to ≤600 mg/day.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have completed the Week 12 Visit in MBX-2H1002 Study.
2. Is an adult ≥18 years of age at the time of the Screening visit of this extension study.
3. Has a diagnosis of one of the following types of hypoparathyroidism for at least 26 weeks prior to the

   Screening visit:
   1. Postsurgical chronic hypoparathyroidism
   2. Idiopathic hypoparathyroidism
   3. Autoimmune hypoparathyroidism
4. Can comprehend and is willing to sign an informed consent form (ICF), and abide by the study restrictions, study visits, and procedures.
5. In the opinion of the investigator, must be able to successfully demonstrate reconstitution and self-administration of study drug.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2027-05-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety and tolerability of weekly MBX 2109 in patients with hypoparathyroidism. | 104 weeks
  Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Locations (22):
- United States (17):
  - MBX Biosciences Investigational Site, Miami, Florida
  - MBX Biosciences Investigational Site, Macon, Georgia
  - MBX Biosciences Investigational Site, Jackson, Mississippi
  - MBX Biosciences Investigational Site, St Louis, Missouri
  - MBX Biosciences Investigational Site, Las Vegas, Nevada
  - MBX Biosciences Investigational Site, Reno, Nevada
  - MBX Biosciences Investigational Site, Albany, New York
  - MBX Biosciences Investigational Site, New York, New York
  - MBX Biosciences Investigational Site, The Bronx, New York
  - MBX Biosciences Investigational Site, Columbus, Ohio
  - MBX Biosciences Investigational Site, Dallas, Texas
  - MBX Biosciences Investigational Site, El Paso, Texas
  - MBX Biosciences Investigational Site, Fort Worth, Texas
  - MBX Biosciences Investigational Site, Round Rock, Texas
  - MBX Biosciences Investigational Site, San Antonio, Texas
  - MBX Biosciences Investigational Site, Weslaco, Texas
  - MBX Biosciences Investigational Site, Madison, Wisconsin
- Argentina (4):
  - MBX Biosciences Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - MBX Biosciences Investigational Site, Córdoba, Río Cuarto
  - MBX Biosciences Investigational Site, Córdoba
  - MBX Biosciences Investigational Site, San Miguel de Tucumán
- MBX Biosciences Investigational Site, Samsun, Turkey (Türkiye)